CLINICAL TRIAL: NCT02008968
Title: Effect of Allopurinol Treatment on Insulin Resistance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Mehmet Kanbay, Associate Professor Doctor Mehmet Kanbay, Istanbul Medeniyet University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Allo2013
Record Dates: First submitted 2013-12-07; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Hyperuricemia; Prediabetes; Insulin Resistance
MeSH Terms: conditions — Hyperuricemia; Prediabetic State; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Uric acid ≥7 mg/dL (Active Comparator): This arm will receive allopurinol treatment. 50 subjects will be recruited.
  Interventions: Drug: allopurinol 300 mg./day
- Uric acid ≥6 and <7 (Active Comparator): This arm will not receive allopurinol. 50 subjects will be recruited.
  Interventions: Other: No intervention
- Normouricemic (Placebo Comparator): This arm is healthy controls. 30 subjects will be recruited.
  Interventions: Drug: Normouricemic

INTERVENTIONS:
Drug: allopurinol 300 mg./day
  Arms: Uric acid ≥7 mg/dL
Other: No intervention
  Arms: Uric acid ≥6 and <7
Drug: Normouricemic
  Arms: Normouricemic

SUMMARY:
Several studies showed that hyperuricemia is an independent risk factor for development of diabetes mellitus. However none of the previous studies have investigated the effect of lowering serum uric acid levels on insulin resistance of which is also named as prediabetes. With this background in mind, we aimed to test the effect of lowering serum uric acid level with allopurinol on insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 30
* Serum uric acid level ≥7mg/dL
* Glomerular filtration rate ≥60 ml/min

Exclusion Criteria:

* presence of Diabetes Mellitus
* history of gout
* history of allopurinol use
* body mass index ≥35 kg/m2
* proteinuria ≥ 1gr/ day
* presence of autoimmune disease
* rheumatology associated disease
* presence of hypothyroidism or hyperthyroidism
* presence of diseases which may cause chronic inflammation or microalbuminuria (e.g. malignancy, chronic liver disease, hypertension, chronic lung disease)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-07 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Change in insulin resistance (HOMA-IR) | baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ali Bakan, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University Goztepe Training and Research Hospital, Istanbul, Marmara, Turkey (Türkiye)